CLINICAL TRIAL: NCT05146752
Title: Application of Schumann Resonance on Premature Infant
Brief Title: The Effect of Schumann Resonance on Preterm Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Hsiao-Ling Chuang, Assistant Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CS19049
Record Dates: First submitted 2021-11-09; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Extremely Low Birth Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extremely low frequency electromagnetic fields (Experimental): After parental permission for participation was obtained, the preterm newborns were enrolled and divided into the experimental group, which received ELF-EMF therapy after a pretest in addition to regular medical care, and the control group, which received regular medical care only, using a random number table.
  Interventions: Device: extremely low frequency electromagnetic fields
- control group (Other): routine care
  Interventions: Other: routine care

INTERVENTIONS:
Device: extremely low frequency electromagnetic fields — extremely low frequency electromagnetic fields
  Arms: Extremely low frequency electromagnetic fields
Other: routine care — routine care
  Arms: control group

SUMMARY:
Body weight gain is crucial for preterm newborns, especially those with a low birth weight. Owing to their noninvasive, noncontact, and non-pharmaceutical properties, extremely low frequency electromagnetic fields (ELF-EMFs) are a promising medium of alternative and complementary therapy.

DETAILED DESCRIPTION:
Sixty-one preterm newborns of 32-35 weeks' gestational age were recruited from the neonatal intensive care unit of the Chung Shan Medical University Hospital and randomly assigned to one of two groups: the experimental group (n = 31) or the control group (n = 30). Both groups received the same medical care, but the experimental group was exposed to ELF-EMFs until discharge.

ELIGIBILITY:
Inclusion Criteria:

* gestational age (GA) between 32 and 35 weeks
* Neonatal Therapeutic Intervention Scoring System (NTISS) score <9

Exclusion Criteria:

* (1) a diagnosis of congenital anomaly, intrauterine growth retardation, cerebral palsy, or hydrocephalus; (2) an NTISS score>9

Ages: 26 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2019-06-08 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-06-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline body weight gain at 4 weeks | Baseline, week1, week2, week3, week4.
  Although the preterm newborns' body weight was recorded daily, the differences in body weight gain between the two groups were compared every week.The body weights of the preterm newborns were recorded using the same weighing scale at the same time every day.

SECONDARY OUTCOMES:
Change from Baseline sleep quality at 4 weeks | Baseline, week1, week2, week3, week4.
  The preterm newborns' sleep quality was recorded daily, the differences in sleep quality between the two groups were compared every week. The preterm' sleep quality was recorded by the sleep tracking devices of Fitbit Alta HR. The correlation coefficient between Alta HR and PSG was 0.85~0.87.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No